CLINICAL TRIAL: NCT05733390
Title: A Phase 2, Randomized, Double-blind, Placebo-Controlled Study to Investigate the Efficacy and Safety of JZP541 in Adults With Irritability Associated With Autism Spectrum Disorder
Brief Title: A Study of JZP541 in Adults With Irritability Associated With Autism Spectrum Disorder
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: A decision has been made to prioritize other pipeline programs and terminate this study.
Sponsor: Jazz Pharmaceuticals (Industry)
Collaborators: GW Research (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JZP541-201; 2022-502355-61-00 (Other: CTIS)
Record Dates: First submitted 2023-02-08; First posted 2023-02-17 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Irritability Associated With Autism Spectrum Disorder; Autism Spectrum Disorder; ASD
Keywords: Irritability; Autism Spectrum Disorder; ASD; JZP541
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- JZP541 (Experimental): Participants who will be randomized to receive JZP541.
  Interventions: Drug: JZP541
- Placebo (Placebo Comparator): Participants who will be randomized to receive placebo.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: JZP541 — Oral suspension
  Arms: JZP541
Other: Placebo — Oral suspension
  Arms: Placebo

SUMMARY:
Behavior dysregulation is commonly associated with people with autism spectrum disorder (ASD). Irritability is a major safety concern in adults with ASD. This study will assess the efficacy and safety of JZP541 in the treatment of adults with irritability associated with ASD.

DETAILED DESCRIPTION:
This randomized, double-blind, placebo-controlled, phase 2 study will evaluate the efficacy and safety of JZP541 in treating irritability in adults with ASD.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 to 45 years inclusive at the time of signing the informed consent
* Has a suitable study partner who keeps in regular contact with the participant, has sufficient knowledge of the participant's behavior to complete the study assessments, able to communicate with site personnel, willing to comply with protocol requirements, and has adequate literacy to complete the protocol-specified questionnaires
* Participant has full scale intelligence quotient (IQ) or General Ability Index (GAI) >45, measured in adulthood using the Wechsler Adult Intelligence Scale - Fourth Edition (WAIS-IV) or Wechsler Adult Intelligence Scale - Second Edition (WASI-II), and the ability to self-report on adverse events (AEs) as determined by the investigator
* Able to cooperate and take part in study assessments, including blood sampling
* Has a current diagnosis of autism spectrum disorder (ASD) as per DSM-5 criteria for ASD [confirmed at screening], which has been confirmed by the Autism Diagnostic Observational Schedule-2nd Edition (ADOS-2) or the Autism Diagnostic Interview-Revised (ADI-R) [lifetime assessment is acceptable]. If no lifetime assessment is available, the ADOS-2 or ADI-R should be performed at screening for diagnosis confirmation
* Has episodes of temper outbursts, aggression, self-injurious behavior or a combination of these issues that interfere with the participant's performance or affect others
* Participant's irritability per Clinical Global Impression of Severity (CGIS) is at least 3 (moderate) at screening and randomization
* All medications taken by the participant that may have an effect on ASD symptoms, behavior, anxiety, or sleep must have been stable for 4 weeks, or 8 weeks for long-acting formulations, prior to the Screening Visit and Visit 2
* Willing to maintain a stable regimen for all participant medications and interventions throughout the study
* Participant is compliant with their current medications
* Male participants must agree to refrain from donating sperm, or be abstinent, or agree to use contraception during the Study Intervention Period and for at least 12 weeks after the last dose of study intervention
* Female participants are eligible if she is not pregnant or breastfeeding as specified
* Women of childbearing potential (WOCBP) must have a negative serum pregnancy test within 14 days before the first dose of study intervention
* Participant (or study partner) is willing and able to give informed consent or assent

Exclusion Criteria:

* Has a severe or profound intellectual disability (ie, IQ or GAI ≤ 45)
* Participant is unable to self-report AEs, as determined by the investigator
* Has a current diagnosis of psychosis spectrum disorders (bipolar disorder with psychotic features, schizo-affective disorder, delusional disorder, or schizophrenia)
* Has a current diagnosis of major depression (participants with depression in remission for at least 12 months may be included)
* Has an established history of psychotic spectrum disorders, early signs of psychosis at screening or Visit 2, or first degree relative with a lifetime diagnosis of psychosis spectrum disorders
* Has had a seizure within the past 2 years
* Has had changes in anticonvulsive therapy within the last 12 weeks
* Has experienced myocardial infarction or clinically significant cardiac dysfunction within the 12 months prior to Visit 1 or has a history of clinically significant arterial vascular disease, including cerebrovascular and cardiovascular disease
* Has supine systolic blood pressure < 90 mmHg or > 150 mmHg or supine diastolic blood pressure < 50 mmHg or > 105 mmHg or a postural drop in systolic blood pressure ≥ 20 mmHg or diastolic blood pressure ≥ 10 mmHg, with or without symptoms, at screening or baseline (prior to randomization)
* Has a QTcF interval > 450 ms or a history of additional risk factors for Torsades de pointes
* Has any other significant disease or disorder which, in the opinion of the investigator, may either put the participant at risk because of participation in the study, may influence the result of the study, or may affect the participant's ability to take part in the study
* Had in the 2 weeks prior to screening or up to randomization any condition that might affect baseline assessments
* Has received administration of strong inducers of CYP3A4 ≤ 14 days prior to first doses of study intervention or have ongoing requirements for these medications
* Is currently using or has used within the 12 weeks prior to screening recreational or medicinal cannabis, cannabinoid-based medications (botanical or synthetic; eg, Sativex, Epidiolex/Epidyolex, Nabilone, Dronabinol) and/or is unwilling to abstain for the duration of the study
* Is currently taking bupropion
* Has received another investigational product within the 12 weeks prior to the Screening Visit
* Has any known or suspected hypersensitivity to cannabinoids or any of the excipients of the study intervention
* Has been previously randomized into this study
* Has impaired liver function at screening, as reflected by serum alanine aminotransferase or aspartate aminotransferase > 1.5 × ULN, or total bilirubin > ULN
* Female participant who is pregnant (positive pregnancy test), lactating, or planning pregnancy during the study or within 3 months thereafter
* Has any history of suicidal behavior or any suicidal ideation (with intent per C-SSRS questions 4 and 5) in the last month at screening (last month) or Visit 2 (randomization)
* Has any known or suspected history of alcohol or substance abuse
* Has positive drug abuse test at screening
* Is living in the same household as another active participant of this study or nominated study partner is actively serving as a study partner for another participant of this study (Note: Same household does not apply to professional care-home environment)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2023-06-30 (Actual); Primary Completion 2023-11-09 (Actual); Study Completion 2023-11-09 (Actual)

PRIMARY OUTCOMES:
Mean Change From Baseline to Week 12 in the Aberrant Behavior Checklist-Irritability (ABC-I) Subscale Score | Baseline to Week 12
  The ABC-I subscale contains 15 items and its score is used to rate a person's irritability over the past 7 days on a 4-point scale, where 0 indicates no irritability and 3 indicates severe irritability. Higher scores indicate worse outcome.

SECONDARY OUTCOMES:
Number of Participants With Treatment-emergent Adverse Events | Day 1 up until end of study or discontinuation (whichever occurs first), up to approximately 2 years
Percentage of Participants with ≥ 25% Reduction in Aberrant Behavior Checklist-Irritability (ABC-I) Subscale Score From Baseline | Baseline up until end of study or discontinuation (whichever occurs first), up to approximately 2 years
  The ABC-I subscale contains 15 items and its score is used to rate a person's irritability over the past 7 days on a 4-point scale, where 0 indicates no irritability and 3 indicates severe irritability. Higher scores indicate worse outcome.
Mean Change in ABC-I Score After Treatment Discontinuation | Date of treatment discontinuation up until end of study or discontinuation (whichever occurs first), up to approximately 2 years
  The ABC-I subscale contains 15 items and its score is used to rate a person's irritability over the past 7 days on a 4-point scale, where 0 indicates no irritability and 3 indicates severe irritability. Higher scores indicate worse outcome.
Mean Change From Baseline in the Caregiver Top 3 ABC-I Items of Concern | Baseline up until end of study or discontinuation (whichever occurs first), up to approximately 2 years
Mean Change From Baseline to Week 12 in Aberrant Behavior Checklist (ABC) Modified Social Withdrawal Subscale Score | Baseline to Week 12
  The ABC Modified Social Withdrawal subscale contains 13 items and its score is used to rate a person's social withdrawal over the past 7 days on a 4-point scale, where 0 indicates no withdrawal and 3 indicates severe/extreme social withdrawal. Higher scores indicate worse outcome.
Mean Change From Baseline to Week 12 in Aberrant Behavior Checklist (ABC) Stereotypic Behavior Subscale Score | Baseline to Week 12
  The ABC Stereotypic Behavior subscale contains 7 items and its score is used to rate a person's stereotypic behavior over the past 7 days on a 4-point scale, where 0 indicates no stereotypic behavior and 3 indicates severe stereotypic behavior. Higher scores indicate worse outcome.
Mean Change From Baseline to Week 12 in Repetitive Behavior Scale - Revised (RBS-R) Subscale Scores | Baseline to Week 12
  The RBS-R subscale score is used to rate a person's behavior over the past 7 days on a 4-point scale, where 0 indicates that the behavior does not occur and 3 indicates that the behavior occurs and is a serious problem. Higher scores indicate worse behavior.

CONTACTS AND LOCATIONS:
Locations (1):
- Albert Einstein College of Medicine, The Bronx, New York, United States